CLINICAL TRIAL: NCT03354962
Title: Induction of Immune-mediated aBscOpal Effect thrOugh STEreotactic Radiation Therapy in Metastatic Melanoma Patients Treated by PD-1 + CTLA-4 Inhibitors (BOOSTER MELANOMA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17 CUTA 11
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
Keywords: Melanoma; Immune checkpoint; Nivolumab; Ipilimumab; Abscopal effect; Stereotactic radiotherapy; PD-1; CTLA-4
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Active Comparator)
  Interventions: Combination Product: Nivolumab + Ipilimumab
- ARM B (Experimental)
  Interventions: Combination Product: Combined treatment schema

INTERVENTIONS:
Combination Product: Nivolumab + Ipilimumab — Nivolumab + Ipilimumab alone (standard dosage regimen)
  Arms: ARM A
Combination Product: Combined treatment schema — SBRT (recommended optimal dose) with Nivolumab + Ipilimumab (standard dosage regimen)
  Arms: ARM B

SUMMARY:
This study is a phase I/II, multicenter, open-label study starting with a phase I part followed by a Phase II part.

The phase I part of the study aims at evaluating the safety and efficacy (in terms of abscopal effect at week 6) of the treatment combination schema of Stereotactic Body Radiation Therapy (SBRT) and PD-1 plus CTLA-4 inhibitors in patients with metastatic melanoma. Patients will be assigned in one of 3 cohorts depending the metastatic site. 18 patients will be enrolled in each cohort.

Once the recommended optimal radiotherapy dose has been declared for the 3 cohorts, patients will be enrolled in the phase II part of the study in order to evaluate the activity (progression-free survival at 6 months) of SBRT given in combination with immune checkpoints inhibitors in patients with metastatic melanoma.

66 patients will be included in the phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-proven metastatic and/or unresectable melanoma (stage IIIc-IV, M1a-c as per AJCC 8th Edition), including mucosal melanoma, without evidence of active intra-cranial disease.
2. Patients with tumor PD-L1 expression <1%.
3. Patients are included regardless of BRAFV600 mutation status. BRAFV600 mutation status must be documented.
4. Patients with a metastatic lesion located on liver, lung, or bone and eligible for a SBRT.
5. Patients should present at least two lesions: one lesion to be irradiated and one distant lesion that will serve as control. Lesion to be irradiated will be selected on the basis of symptomatology, safety and/or location. Preferentially, both lesions should be measurable per RECIST 1.1. If only the control lesion is measurable but not the irradiated lesion, eligibility will be discussed with the sponsor.
6. Age ≥18 years at the time of study entry.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
8. Life expectancy of at least 3 months.
9. Patients able to participate and willing to give informed consent prior to performance of any study-related procedures and to comply with the study protocol.
10. Screening laboratory values must meet the following criteria and should be obtained prior to commencement of treatment:

    * White blood count (WBC) ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Hemoglobin > 9.0 g/dL
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula)
    * AST/ALT ≤ 3 x ULN (except subjects with hepatic metastasis, who can have AST/ALT ≤ 5 x ULN)
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
11. Adequate cardiac and respiratory functions defined as New York Heart Association (NYHA) class 1 and SaO2 > 90%.
12. Patient must be naïve to systemic treatment for locally advanced and/or metastatic disease (i.e., no prior systemic anticancer therapy for advanced disease; stage IIIc and IV). Prior adjuvant therapies (including Interferon α and Ipilimumab) is permitted if it was completed at least 12 weeks before start of treatment and all related AEs have either returned to baseline or stabilized.
13. Prior radiotherapy or radiosurgery must have been completed at least 4 weeks prior to the first dose of the study treatment.
14. Women of childbearing potential (WOCBP) must use two appropriate methods of contraception to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab/Ipilimumab to undergo five half-lives) after the last dose of investigational drug.
15. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
16. Men who are sexually active with WOCBP must use two contraceptive methods including at least one method with a failure rate of less than 1% per year for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception
17. Absence of any psychological, familial, sociological or geographical condition that potentially hampers compliance with the study protocol and follow-up after treatment discontinuation schedule.
18. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patient pregnant, or breast-feeding.
2. Uveal melanoma.
3. Active and/or symptomatic intra cranial metastasis (including melanomatous meningitis).
4. Previous treatment with B-RAF or MEK inhibitors within 12 weeks prior start of treatment.
5. Hypersensitivity to the drugs of the study.
6. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Clinically significant cardiac dysfunction including congenital, familial, and genetic cardiac disorders, current instable angina, current symptomatic congestive heart failure of NYHA class 2 and higher, current uncontrolled hypertension ≥ grade 3; Left Ventricular Ejection Fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower.
8. Patient with active malignancy other than melanoma or a history of previous within the past 3 years; except for patients with resected Basal cell carcinoma or resected Spindle cell carcinoma, resected carcinoma in situ of the cervix and resected carcinoma in situ of the breast.
9. Active, known or suspected autoimmune disease including but not restricted to multiple sclerosis, optical nevritis and demyelinating neuropathy. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
10. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (ribonucleic acid or HCV antibody) indicating acute or chronic infection.
11. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
12. Vaccination with any live attenuated conventional vaccine within the 3 months preceding the start of study treatment.
13. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection.
14. Patient included in another study with an experimental molecule and/or procedure.
15. Unwillingness or inability to provide written informed consent.
16. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the compliance of treatment and the study protocol.
17. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose Limiting Toxicities (DLT) incidence. | 3 weeks per patient
Phase I: Abscopal effect. | 6 weeks per patient
  Abscopal effect is defined as a tumor shrinkage ≥ 20% compared to baseline in the control lesion (non-irradiated and distant lesion) at the end of the 6-week period of treatment without evidence of clinical progression.
Phase II: The primary endpoint is the rate of patients alive without progression at 6 months. | 6 months per patient

SECONDARY OUTCOMES:
Phase I: Safety will be evaluated using NCI CTCAE V4.03 criteria. | 15 months per patient
Phase II: Progression Free Survival (PFS) is defined as the time from inclusion until progression or death. | 24 months per patient
Phase II: Safety will be evaluated using NCI CTCAE V4.03. | 15 months per patient
Phase II: Pattern of response rate will be followed in irradiated and non-irradiated lesions separately by CT-scan evaluation using RECIST V1.1. | 24 months per patient

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Chu Bordeaux, Bordeaux
  - Centre Oscar Lambret, Lille
  - ICM, Montpellier
  - CHU NICE, Nice
  - Centre Eugene Marquis, Rennes
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse